CLINICAL TRIAL: NCT03913455
Title: A Phase II Study Evaluating Efficacy and Safety of Hypomethylating Agent Guadecitabine in Combination With Carboplatin in Extensive Stage Small Cell Lung Cancer
Brief Title: Guadecitabine in Combination With Carboplatin in Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shadia Jalal, MD (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry); Indiana University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Shadia Jalal, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN LUN17-302
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Small Cell Lung Cancer; Extensive-stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — guadecitabine; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Guadecitabine and Carboplatin (Other): Each cycle = 28 days; Subjects receive 4 cycles
  Interventions: Drug: Guadecitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Guadecitabine — Guadecitabine 30 mg/m2 subcutaneously Days 1-5
  Other Names: SGI-110
Drug: Carboplatin — Carboplatin AUC 4 IV Day 5
  Other Names: Platinol

SUMMARY:
This is a phase II, open-label, single arm, single-stage study. Both, chemo-sensitive and chemo-resistant patients will be enrolled and treated with 4 cycles of combination of Guadecitabine and carboplatin

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age ≥ 18 years.
* Histological or cytological diagnosis of small cell lung cancer. Subjects must have extensive-stage disease is defined as disease beyond the ipsilateral hemithorax, mediastinum and ipsilateral supraclavicular area and including malignant pleural or pericardial effusion or hematogenous metastases.
* Patient should not have received more than 1 prior line of chemotherapy (could have received immunotherapy which does not count as chemotherapy).
* ECOG PS 0-1
* Measurable disease as per RECIST v1.1. Subjects may have bone-only disease. NOTE: Bone-only subjects are eligible if their disease can be documented/evaluated by bone scans, CT or MRI. Their disease will be assessed using MD Anderson criteria. NOTE: Previously irradiated lesions are eligible as a target lesion only if there is documented progression of the lesion after irradiation.
* Adequate bone marrow, liver, and renal function, as assessed by the following laboratory requirements:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Platelet count ≥ 100,000/mm3
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN). For subjects with Gilbert's Disease, total bilirubin ≤ 3 x ULN
  * ALT and AST ≤ 2.5 x ULN. For subjects with documented liver metastases, ALT and AST ≤ 5×ULN
  * International Normalized Ratio (INR) ≤1.5, if not therapeutically anticoagulated. Subjects who are being therapeutically anticoagulated may be included provided that the anticoagulation regimen is stable and closely monitored.
  * Estimated glomerular filtration rate (eGFR) ≥ 60 mL/minute/1.73 m2 as determined using the Cockcroft-Gault formula.
* Women of child-bearing potential must not be pregnant or breastfeeding and must have a negative pregnancy test at screening.
* Male and female subjects of child- bearing potential must agree to use an effective method of birth control from the screening visit through 6 months after the last dose of study drug.

Exclusion Criteria:

* Platinum refractory disease defined as disease progression during first line platinum containing chemotherapy regimen. Progression following platinum based therapy is allowed.
* Prior therapy with a hypomethylating agent.
* Previously untreated (non-irradiated), symptomatic brain metastases. No prior treatment is required for non-symptomatic brain metastases. Previously treated symptomatic brain metastases are permitted.
* Unstable or clinically significant concurrent medical condition, psychiatric illness or social situation that would, in the opinion of the investigator, jeopardize the safety of a subject and/or their compliance with the protocol.
* Clinically significant acute infection requiring systemic antibacterial, antifungal, or antiviral therapy. (Suppressive therapy for chronic infections allowed, for example: Subjects with HIV/AIDS with adequate antiviral therapy to control viral load would be allowed. Subjects with viral hepatitis with controlled viral load would be allowed while on suppressive antiviral therapy.)
* Hypersensitivity to (IMP) or components of the study treatment regimen.
* Treated with any investigational drug within 3 weeks of first dose of study treatment.
* Pregnant or breastfeeding.
* Second malignancy currently requiring active therapy except breast or prostate cancer stable on or responding to endocrine therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2022-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shadia Jalal, MD, MBBS, Principal Investigator — Indiana University School of Medicine
Locations (4):
- United States (4):
  - Indiana Univeristy Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Ball Memorial Cancer Center, Muncie, Indiana
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Wisconsin, Clinical Cancer Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Guadecitabine and Carboplatin
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Guadecitabine and Carboplatin
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 62.5 [43 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Smoking Status [Count of Participants; unit: Participants]
  Current | 10
  Former | 13
  Never | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD. PFS is defined as time from registration until disease progression met by RECIST 1.1 or death from any cause.
Time Frame: Time of treatment start until the criteria for disease progression or death. Up to a maximum of 7 months.
Population: Out of 24 subjects, 15 subjects were in Platinum Sensitive group and 9 subjects were in Platinum Resistant group.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Guadecitabine and Carboplatin (Platinum Sensitive); Guadecitabine and Carboplatin (Platinum Resistant): Each cycle = 28 days; Subjects receive 4 cycles
  Guadecitabine: Guadecitabine 30 mg/m2 subcutaneously Days 1-5
  Carboplatin: Carboplatin AUC 4 IV Day 5
Arm/Group | Guadecitabine and Carboplatin (Platinum Sensitive) | Guadecitabine and Carboplatin (Platinum Resistant)
Number analyzed (Participants) | 15 | 9
Months | 1.9 [1.2 to 2.5] | 1.7 [0.9 to 4.1]

2. Secondary Outcome: Adverse Events
Description: All adverse events (AEs) had been determined according to the NCI Common Terminology Criteria for (NCI CTCAE) V5. A summary of the total number of participants is provided.
Time Frame: AEs had been recorded from time of signed informed consent until 30 days after discontinuation of study drug(s) or until a new anti-cancer treatment starts, whichever occurs first, up to a maximum of 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Guadecitabine and Carboplatin
Number analyzed (Participants) | 24
Participants | 24

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  ORR is defined as the proportion of all subjects with confirmed PR or CR according to RECIST 1.1
Time Frame: Up to a maximum of 7 months
Population: Out of 24 subjects, 15 subjects were in Platinum Sensitive group and 9 subjects were in Platinum Resistant group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Guadecitabine and Carboplatin (Platinum Sensitive) | Guadecitabine and Carboplatin (Platinum Resistant)
Number analyzed (Participants) | 15 | 9
Percentage of participants | 7.1 [0.2 to 33.9] | 0 [NA to NA] — No patients on Platinum Resistant group achieved confirmed CR or PR.

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  DCR defined as CR + PR + Stable Disease (SD) >=8 weeks per RECIST 1.1
Time Frame: Up to a maximum of 7 months
Population: Out of 24 subjects, 15 subjects were in Platinum Sensitive group and 9 subjects were in Platinum Resistant group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Guadecitabine and Carboplatin (Platinum Sensitive) | Guadecitabine and Carboplatin (Platinum Resistant)
Number analyzed (Participants) | 15 | 9
Percentage of participants | 42.9 [17.7 to 71.1] | 33.3 [7.5 to 70.1]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from treatment start until death or date of last contact.
Time Frame: Time of treatment start until death or date of last contact, up to a maximum of 16 months.
Population: Out of 24 subjects, 15 subjects were in Platinum Sensitive group and 9 subjects were in Platinum Resistant group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Guadecitabine and Carboplatin (Platinum Sensitive) | Guadecitabine and Carboplatin (Platinum Resistant)
Number analyzed (Participants) | 15 | 9
Months | 6.8 [2.7 to 10] | 4.4 [1.4 to 11.4]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 16 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored for up to 5 months.
Arm/Group | Guadecitabine and Carboplatin
All-Cause Mortality (participants affected / at risk) | 18/24
Serious Adverse Events (participants affected / at risk) | 6/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guadecitabine and Carboplatin (N=24)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
LOWER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
SEPSIS (Infections and infestations) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guadecitabine and Carboplatin (N=24)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (8)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 (2)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (3)
ANEMIA (Blood and lymphatic system disorders) | 12 (15)
ANOREXIA (Metabolism and nutrition disorders) | 6 (7)
ANXIETY (Psychiatric disorders) | 3 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 5 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (6)
BELCHING (Gastrointestinal disorders) | 1 (1)
BLOATING (Gastrointestinal disorders) | 1 (1)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
BLOOD PROLACTIN ABNORMAL (Investigations) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
COLONIC ULCER (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 8 (8)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (4)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (2)
DIARRHEA (Gastrointestinal disorders) | 5 (5)
DRY MOUTH (Gastrointestinal disorders) | 2 (2)
DYSGEUSIA (Nervous system disorders) | 5 (7)
DYSPHAGIA (Gastrointestinal disorders) | 2 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 7 (8)
DYSURIA (Renal and urinary disorders) | 1 (1)
EAR AND LABYRINTH DISORDERS - OTHER, SPECIFY (Ear and labyrinth disorders) | 1 (1)
EDEMA LIMBS (General disorders) | 3 (3)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 1 (1)
ESOPHAGEAL PAIN (Gastrointestinal disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 3 (3)
FATIGUE (General disorders) | 14 (20)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
FEVER (General disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 1 (2)
HEADACHE (Nervous system disorders) | 3 (4)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (2)
HOT FLASHES (Vascular disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPERLIPIDEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (3)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 6 (9)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (3)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPONATREMIA (Metabolism and nutrition disorders) | 4 (5)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPOTENSION (Vascular disorders) | 2 (3)
INJECTION SITE REACTION (General disorders) | 6 (11)
INSOMNIA (Psychiatric disorders) | 5 (6)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 (2)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 1 (1)
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 10 (24)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 10 (14)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
PAIN (General disorders) | 7 (16)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (4)
PARESTHESIA (Nervous system disorders) | 2 (2)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (4)
PLATELET COUNT DECREASED (Investigations) | 4 (5)
PRESYNCOPE (Nervous system disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1)
SINUS PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 2 (2)
SKIN INFECTION (Infections and infestations) | 2 (3)
TESTOSTERONE DEFICIENCY (Endocrine disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
THRUSH (Infections and infestations) | 2 (2)
TOOTH INFECTION (Infections and infestations) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2)
VAGINAL INFECTION (Infections and infestations) | 1 (1)
VOMITING (Gastrointestinal disorders) | 6 (8)
WEIGHT GAIN (Investigations) | 1 (1)
WEIGHT LOSS (Investigations) | 5 (6)
WHITE BLOOD CELL DECREASED (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT03913455/Prot_SAP_000.pdf